CLINICAL TRIAL: NCT01946945
Title: Comparison of Standard ART Practice vs. Trophectoderm Biopsy, Whole Chromosome Analysis by Next Generation Sequencing, and Replacement of a Single Euploid Embryo
Brief Title: Comparison of Standard ART Practice vs. Trophectoderm Biopsy and Whole Chromosome Analysis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Reprogenetics (Industry)
Collaborators: Main Line Fertility Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: Reprogenetics-3.109
Record Dates: First submitted 2013-08-27; First posted 2013-09-20 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Infertility; Recurrent Pregnancy Loss
Keywords: infertility; recurrent pregnancy loss; miscarriage; Next Generation Sequencing
MeSH Terms: conditions — Infertility; Abortion, Spontaneous

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control - Standard ART treatment (No Intervention)
- Test - PGS (Experimental): All embryos will be hatched on day 3. Patients will have hatching blastocysts (*) biopsied on day 5,/6. Embryos will be vitrified. Patients will have a single hatching euploid blastocyst (*) replaced on a thawed cycle.
  Interventions: Genetic: Next Generation Sequencing after Blastocyst biopsy

INTERVENTIONS:
Genetic: Next Generation Sequencing after Blastocyst biopsy — PGD using blastocyst biopsy and testing of the biopsy by NGS
  Other Names: PGD: Preimplantation Genetic Diagnosis
  Arms: Test - PGS

SUMMARY:
We propose to perform a clinical randomized trial to evaluate the effect of blastocyst biopsy and whole chromosome analysis by Next Generation Sequencing (NGS) in comparison to standard Assisted Reproductive Technologies (ART) methods on on implantation rates, miscarriage rates, and pregnancy rates.

This will be three studies into one: a) a comparison of treatment (NGS) and no treatment, b) a non-selection study based on the control group for which we will replace without knowing the ploidy of the embryos, but we will know it later, c) a retrospective study about the use of Mitochondrial DNA as a selection tool.

DETAILED DESCRIPTION:
Patients following the inclusion criteria will be randomized into two groups:

1. Control group: All blastocyst embryos will be biopsied on day 5/6, but the biopsies will be frozen and will not be analyzed before replacement. Blastocyst embryos will be vitrified for future frozen embryo transfer (FET) cycle. Patients will have a single hatching blastocyst (*) thawed and transferred into the uterus in a FET cycle based on standard embryo quality assessment without NGS. After transfer, all biopsied samples will be analyzed (the replaced embryo also, in order to do a non-selection study). If patients in the control group do not have a pregnancy to term from that FET cycle, euploid frozen blastocysts will be thawed and transferred on the next FET transfer.
2. Test group: All blastocyst embryos will be biopsied on day 5/6, and the biopsies will be analyzed using NGS. (*) and Biopsied blastocyst embryos will be vitrified for a future frozen embryo transfer (FET) cycle. Patients will have a single hatching euploid blastocyst (*) thawed and transferred into the uterus in a FET cycle

(*) Hatching blastocysts as described by Gardner and Schoolcraft (1999)

The Primary efficacy endpoint of comparing the study group with the control will be ongoing implantation rate (# fetus reaching 2nd trimester / # embryos replaced).

All biopsied embryos from the test and control group will have their mitochondrial DNA analyzed, but that information will not be used for purposes of choosing embryos for replacement. Retrospectively but blindly (see blinding of results section), the information will be used at the end of the study to determine which embryos have a higher chance of implanting. If at that point the participating patients have remaining embryos frozen, they will be able to use that information for purposes of embryo selection.

ELIGIBILITY:
Inclusion Criteria:

* All patients medically cleared to do a fresh or frozen embryo transfer.
* Age up to 42 years

Exclusion Criteria:

* microsurgical epididymal sperm aspiration (MESA) and Testicular sperm extraction (TESE) patients
* At least one partner carrier of a chromosomal or genetic disease
* Abnormal ovarian reserve, defined as follicle stimulating hormone (FSH) of >10 IU/L on day 2-4 of the cycle and anti-mullerian hormone (AMH) < 1ng /ml (If only one of the two parameters altered then patients is acceptable). This is based on Mandy Katz abstract at American Society for Reproductive Medicine (ASRM) 2011 where they showed that these patients have 35% chance of having no euploid embryos - They are excluded only to make the study size smaller, otherwise, if an euploid embryo is found in these patients, they implant as well as patients with normal ovarian reserve. Not all centers do AMH testing - we recommend first to run FSH and only test AMH if FSH is abnormal.
* Egg donor cycle (sperm donor is acceptable)
* Gender selection cycles
* Thaw cycles

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
improvement in ongoing implantation rates | When a fetal heartbeat is detected for each patient. (8 weeks after implantation).
  We foresee a significant increase in ongoing implantation rates in the Test group compared to the Control group based on several studies showing about a 50% improvement of implantation rates after Preimplantation Genetic Diagnosis (PGD) with blastocyst biopsy and comprehensive chromosome analysis techniques The center participating in the study has an average 41.5% implantation rate of blastocysts in patients 35-39 years of age without PGD. Assuming that NGS will increase the detection power of chromosome abnormalities, we expect a higher implantation rate in the test group.
  Furthermore, we expect a 6% miscarriage rate in the Test group, based on extensive data from array comparative genomic hybridization (aCGH) results (Hodes-Wertz et al. 2012), while about 21% in the Control group based on Society for Assisted Reproductive Technologies (SART) data (ages 35-40, SART 2011).

SECONDARY OUTCOMES:
Determine specificity and sensitivity rates | During a pregnancy term
  The pregnancy outcome of Controls patients with euploid embryos replaced will be compared to that of control patients with aneuploid embryos replaced. This will give us the specificity of the test (false positive rate) by obtaining the ongoing pregnancy rate of cycles with aneuploid embryos replaced, and the sensitivity of the test (false negative rate) by obtaining the miscarriage rate and ongoing pregnancy rate of cycles with euploid embryos replaced.

OTHER OUTCOMES:
Correlation of Mitochondrial DNA and implantation | When a fetal heartbeat is detected (8 weeks after implantation)
  The third aim of this study is to determine retrospectively if mt DNA content is linked to implantation potential and if that is measurable by NGS. NGS provides the additional advantage that it can measure mitochondrial DNA, which it's content, seems to be inversely correlated with implantation (Fragouli et al 2013, ASRM).

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Munne, PhD, Study Director — Reprogenetics
Locations (1):
- Reprogenetics, Livingston, New Jersey, United States

REFERENCES:
- [Background] Cohen J, Wells D, Munne S. Removal of 2 cells from cleavage stage embryos is likely to reduce the efficacy of chromosomal tests that are used to enhance implantation rates. Fertil Steril. 2007 Mar;87(3):496-503. doi: 10.1016/j.fertnstert.2006.07.1516. Epub 2006 Dec 4. PMID 17141767
- [Background] De Vos A, Staessen C, De Rycke M, Verpoest W, Haentjens P, Devroey P, Liebaers I, Van de Velde H. Impact of cleavage-stage embryo biopsy in view of PGD on human blastocyst implantation: a prospective cohort of single embryo transfers. Hum Reprod. 2009 Dec;24(12):2988-96. doi: 10.1093/humrep/dep251. Epub 2009 Sep 21. PMID 19773223
- [Background] Gutierrez-Mateo C, Colls P, Sanchez-Garcia J, Escudero T, Prates R, Ketterson K, Wells D, Munne S. Validation of microarray comparative genomic hybridization for comprehensive chromosome analysis of embryos. Fertil Steril. 2011 Mar 1;95(3):953-8. doi: 10.1016/j.fertnstert.2010.09.010. Epub 2010 Oct 25. PMID 20971462
- [Background] Munne S, Wells D, Cohen J. Technology requirements for preimplantation genetic diagnosis to improve assisted reproduction outcomes. Fertil Steril. 2010 Jul;94(2):408-30. doi: 10.1016/j.fertnstert.2009.02.091. Epub 2009 May 5. PMID 19409550
- [Background] Schoolcraft WB, Fragouli E, Stevens J, Munne S, Katz-Jaffe MG, Wells D. Clinical application of comprehensive chromosomal screening at the blastocyst stage. Fertil Steril. 2010 Oct;94(5):1700-6. doi: 10.1016/j.fertnstert.2009.10.015. Epub 2009 Nov 25. PMID 19939370
- [Background] Ata B, Kaplan B, Danzer H, Glassner M, Opsahl M, Tan SL, Munne S. Array CGH analysis shows that aneuploidy is not related to the number of embryos generated. Reprod Biomed Online. 2012 Jun;24(6):614-20. doi: 10.1016/j.rbmo.2012.02.009. Epub 2012 Feb 25. PMID 22503277
- [Background] Cohen J, DeVane GW, Elsner CW, Kort HI, Massey JB, Norbury SE. Cryopreserved zygotes and embryos and endocrinologic factors in the replacement cycle. Fertil Steril. 1988 Jul;50(1):61-7. doi: 10.1016/s0015-0282(16)60009-2. PMID 3384119
- [Background] Forman EJ, Hong KH, Ferry KM, Tao X, Taylor D, Levy B, Treff NR, Scott RT Jr. In vitro fertilization with single euploid blastocyst transfer: a randomized controlled trial. Fertil Steril. 2013 Jul;100(1):100-7.e1. doi: 10.1016/j.fertnstert.2013.02.056. Epub 2013 Mar 30. PMID 23548942
- [Background] Fragouli E, Spath K, Alfarawati S, Wells D (2013) Quantification of mitochondrial DNA predicts the implantation potential of chromosomally normal embryos. Fertil Steril, in press (ASRM abstract)
- [Background] Gardner DK and Schoolcraft WB. In vitro culture of human blastocysts. In: Jansen R, Mortimer D. eds. Towards Reproductive Certainty: Fertility and Genetics Beyond 1999. Carnforth, Parthenon Publishin, 1999, 378-88
- [Background] Hodes-Wertz B, Grifo J, Ghadir S, Kaplan B, Laskin CA, Glassner M, Munne S. Idiopathic recurrent miscarriage is caused mostly by aneuploid embryos. Fertil Steril. 2012 Sep;98(3):675-80. doi: 10.1016/j.fertnstert.2012.05.025. Epub 2012 Jun 7. PMID 22683012
- [Background] SART (2011): https://www.sartcorsonline.com/rptCSR_PublicMultYear.aspx?ClinicPKID=0
- [Background] Scott RT Jr, Ferry K, Su J, Tao X, Scott K, Treff NR. Comprehensive chromosome screening is highly predictive of the reproductive potential of human embryos: a prospective, blinded, nonselection study. Fertil Steril. 2012 Apr;97(4):870-5. doi: 10.1016/j.fertnstert.2012.01.104. Epub 2012 Feb 2. PMID 22305103
- [Background] Treff NR, Su J, Tao X, Levy B, Scott RT Jr. Accurate single cell 24 chromosome aneuploidy screening using whole genome amplification and single nucleotide polymorphism microarrays. Fertil Steril. 2010 Nov;94(6):2017-21. doi: 10.1016/j.fertnstert.2010.01.052. Epub 2010 Feb 26. PMID 20188357
- [Background] Treff NR, Ferry KM, Zhao T, Su J, Forman EJ, Scott RT (2011) Cleavage stage embryo biopsy significantly impairs embryonic reproductive potential while blasto- cyst biopsy does not: a novel paired analysis of cotransferred biopsied and non-biopsied sibling embryos. Fertil Steril, 96: Supplement, S2
- [Background] Wells W, Kaur K, Fragouli E, Munné S (2013) Next generation sequencing. Reprod Biomed Online 26: Suppl 1, 55.
- [Background] Yang Z, Liu J, Collins GS, Salem SA, Liu X, Lyle SS, Peck AC, Sills ES, Salem RD. Selection of single blastocysts for fresh transfer via standard morphology assessment alone and with array CGH for good prognosis IVF patients: results from a randomized pilot study. Mol Cytogenet. 2012 May 2;5(1):24. doi: 10.1186/1755-8166-5-24. PMID 22551456
- [Derived] Cornelisse S, Zagers M, Kostova E, Fleischer K, van Wely M, Mastenbroek S. Preimplantation genetic testing for aneuploidies (abnormal number of chromosomes) in in vitro fertilisation. Cochrane Database Syst Rev. 2020 Sep 8;9(9):CD005291. doi: 10.1002/14651858.CD005291.pub3. PMID 32898291